CLINICAL TRIAL: NCT07168356
Title: A Phase 1, Open-Label, Single-Dose, Parallel Group, 2-Part Study to Evaluate the Pharmacokinetics of Bepirovirsen in Adult Participants With Severe or Moderate Renal Impairment Compared to Matched Healthy Control Participants
Brief Title: A Study to Evaluate Blood Levels of Bepirovirsen in Adult Participants With Severe or Moderate Kidney Disease
Acronym: B-Kind
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205872
Record Dates: First submitted 2025-09-10; First posted 2025-09-11 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Hepatitis B
Keywords: Bepirovirsen; Pharmacokinetics; Severe renal impairment; Moderate renal impairment; Healthy participants; Renal function; Kidney disease; Hepatitis B
MeSH Terms: conditions — Hepatitis B; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1- Severe Renal Impairment Participants (Experimental): Participants with severe renal impairment will receive Bepirovirsen.
  Interventions: Drug: Bepirovirsen
- Group 2- Moderate Renal Impairment Participants (Experimental): Participants with moderate renal impairment will receive Bepirovirsen.
  Interventions: Drug: Bepirovirsen
- Group 3-Healthy Control Participants (Experimental): Healthy control participants will receive Bepirovirsen.
  Interventions: Drug: Bepirovirsen

INTERVENTIONS:
Drug: Bepirovirsen — Bepirovirsen will be administered.

SUMMARY:
This is a 2-part study where all participants will receive bepirovirsen. The study will measure how much bepirovirsen from a single dose gets into the blood, and how long it stays in the blood. The purpose of the study is to understand if blood levels of bepirovirsen are different in adults with kidney disease compared to healthy adults who do not have kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, inclusive
* Body weight greater than or equal to 50 kilograms (kg) and body mass index (BMI) within the range 19 to 40 kilograms per square meter (kg/m^2).
* Males and females may participate. Female participants must not be pregnant or breastfeeding, and must be of non-childbearing potential, or agree to use a highly effective method of contraception.
* Capable of giving signed informed consent Additional inclusion criteria for renal impairment groups (Group 1 and Group 2)
* Severe renal impairment [estimated glomerular filtration rate (eGFR) adjusted for actual body surface area (BSA) less than 30 milliliters per minute (ml/min); Group 1] or moderate renal impairment [eGFR adjusted for actual BSA between 30 and 59 ml/min; Group 2], from any cause other than vasculitis or glomerulonephritis Additional inclusion criteria for healthy control participants with normal renal function (Group 3)
* Healthy, based on medical evaluation including medical history, physical examination, laboratory tests, and electrocardiogram (ECG).
* Normal renal function (eGFR adjusted for actual BSA greater than or equal to 90 ml/min)

Exclusion Criteria:

* Any medical condition that could affect the absorption, metabolism, or elimination of drugs, increase the risk of taking part in the study, or interfere with interpretation of the study data.
* History of vasculitis or any type of glomerulonephritis
* Use of creatine-containing supplements within 30 days of screening or intended use during the study.
* Current enrolment in another interventional study, or past participation in a study where an investigational medicine, vaccine or device was administered if, at the time of consent, it is within 5 half-lives or twice the duration of the biological effect (whichever is longer) of the product given in the previous study.
* Received any oligonucleotide or small interfering ribonucleic acid (siRNA) within the past 12 months.
* Exposure to more than 4 investigational products within the past 12 months.
* A positive blood test for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Average weekly alcohol intake of greater than 14 drinks for males or greater than 7 drinks for females.
* Current substance misuse or dependence, or a previous history of substance misuse or dependence that could interfere with ability to participate in the study.

Additional exclusion criteria for renal impairment groups (Group 1 and Group 2)

* History of renal transplantation or anticipated renal transplant during the study.
* On dialysis or likely to require dialysis during the study.
* Positive drug or alcohol screen (unless because of prescribed medication). Additional exclusion criterion for healthy control group (Group 3)
* Positive drug or alcohol screen.
* Urine albumin-to-creatinine ratio (uACR) > 0.3 mg/mg (300 mg/g).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-04-28 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Plasma Area Under the Concentration Time Curve From Time Zero (Pre-Dose) Extrapolated to Infinite Time [AUC(0-∞)] of Bepirovirsen | Up to Day 50
Maximum Observed Concentration (Cmax) of Bepirovirsen | Up to Day 50

SECONDARY OUTCOMES:
Plasma Area Under the Concentration Time Curve From Time Zero (Pre-Dose) to 24 hours [AUC(0-24)] of Bepirovirsen | Up to 24 hours
Plasma Area Under the Concentration Time Curve From Time Zero (Pre-Dose) to 168 hours (Day 8) [AUC(0-168)] of Bepirovirsen | Up to 168 hours
Observed Concentration of Bepirovirsen on Day 8 | At Day 8
Apparent Terminal Phase Half-life (t1/2) of Bepirovirsen | Up to Day 50
Apparent Clearance (CL/F) of Bepirovirsen | Up to Day 50
Time of Occurrence of Cmax (Tmax) of Bepirovirsen | Up to Day 50
Apparent Terminal Phase Volume of Distribution (Vz/F) of Bepirovirsen | Up to Day 50

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf